CLINICAL TRIAL: NCT03681990
Title: Evaluation of Microbial Population Reductions Within a Defined Product Coverage Area
Brief Title: In Vivo Preoperative Skin Preparation Efficacy Study Within a Defined Product Coverage Area
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EM-012926
Record Dates: First submitted 2017-07-31; First posted 2018-09-24 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Surgical Skin Preparation; Surgical Procedure, Unspecified
Keywords: surgical skin prep; CHG; IPA
MeSH Terms: interventions — Chromogranins; chlorhexidine gluconate; Ethanol; 2-Propanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 3M CHG/IPA Prep / Center (Experimental): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; sample collected from center test site on skin in application area.
  Interventions: Drug: 3M CHG/IPA Prep
- 3M CHG/IPA Prep / Mid-peripheral (Experimental): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; sample collected from mid-peripheral test site on skin in application area.
  Interventions: Drug: 3M CHG/IPA Prep
- 3M CHG/IPA Prep / Peripheral (Experimental): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; sample collected from peripheral test site on skin in application area.
  Interventions: Drug: 3M CHG/IPA Prep

INTERVENTIONS:
Drug: 3M CHG/IPA Prep — Apply topically to intact skin
  Other Names: CHG 2%/IPA 70%; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%; Chlorhexidine gluconate and Isopropyl alcohol

SUMMARY:
This study evaluates reduction of resident flora produced by the test product within a defined prepped area of skin.

DETAILED DESCRIPTION:
Three different sample sites within a defined prepped area of skin were collected to determine whether reductions in resident flora produced by the test product are consistent.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects of any race who are at least 18 years of age,
* Subjects must have an area on their back region to accommodate the treatment coverage area,
* Subjects must be in good general health,
* Subjects who satisfy all inclusion/exclusion criteria and will voluntarily read and sign the Informed Consent Form,
* Subjects who have good skin condition on the test sites,
* Subjects who are willing to report to the study facility approximately 72 hours prior to Screening or Treatment Day for clipping, if needed,
* Subjects who are willing to avoid showering and tub-bathing within 72 hours prior to Screening and Treatment Days, and
* Subjects who have Screening Day baseline counts of > 3.00 log10 per cm2 in each of the 3 sample sites (center, mid-peripheral and peripheral) in the treatment area (back region).

Exclusion Criteria:

* Participation in another clinical study in the past 30 days, current participation in another clinical study, or previous participation in this study,
* Has taken antihistamines in the 48 hours prior to Treatment Day,
* Any tattoos, scars, breaks in the skin, or any form of dermatitis, or other skin disorders (including acne) on the applicable test areas,
* A history of skin allergies,
* A history of skin cancer within 6 inches of the test areas,
* Known sensitivity to acrylate-, chlorhexidine gluconate-, or alcohol-containing products, or to medical tape, metals, natural rubber latex, vinyl, or skin-marking inks,
* A medical diagnosis with physical condition that may put the subject at risk, such as a current or recent severe illness, hepatitis, organ transplant, congestive heart disease, or any immunocompromised conditions, such as AIDS (or HIV positive),
* Any medical condition or use of any medications that, in the opinion of the Investigator, should preclude participation,
* Topical antimicrobial exposure within 14 days prior to Screening Day and throughout the study. Restrictions include, but are not limited to antimicrobial soaps, medicated shampoos, medicated lotions, antiperspirants/deodorants, perfumes, after shaves, and colognes,
* Use of systemic or topical antibiotic medications, steroid medications, or any other product known to affect the normal microbial flora of the skin within 14 days prior to Screening Day and throughout the study,
* Exposure of the test areas to solvents, acids, bases, strong detergents, fabric softener-treated clothing, or other household chemicals within 14 days prior to Screening Day and throughout the study,
* Swimming in chemically treated pools or bathing in hot tubs, spas, or whirlpools within 14 days prior to Screening Day and throughout the study,
* Use of tanning beds, hot waxes, or depilatories (in the applicable test areas) within 14 days prior to Screening Day and throughout the study
* Bathing and showering within 72 hours prior to Screening Day and throughout the study, or
* Subject has used moisturizers or any topical treatment (e.g. lotion, sunscreen or shaving cream) on the test sites in the 24-hour period prior to Screening Day and Treatment Day participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozalia Olsavszky, MD, Principal Investigator — Eurofins/Evic
Locations (1):
- Eurofins Evic Romania/S.C. BIO HIGH TECH S.R.L., Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG/IPA Prep: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; samples collected from center, mid-periphery, and periphery of test site on skin in application area.
Period: Overall Study
Arm/Group | 3M CHG/IPA Prep
Started | 28; 84 test sites on skin
Completed | 28; 84 test sites on skin
Not Completed | 0; 0 test sites on skin

BASELINE CHARACTERISTICS:
Arm/Group | 3M CHG/IPA Prep / Center
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 4
Sex/Gender, Customized [Number; unit: participants]
  Female | 0
  Male | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Ethnicity - Hispanic or Latino | 0
  Ethnicity - Not Hispanic or Latino | 28
  Race - American Indian or Alaska Native | 0
  Race - Asian | 0
  Race - Native Hawaiian or Other Pacific Islander | 0
  Race - Black or African American | 0
  Race - White | 28
  Race - More than one race | 0
  Race - Unknown or not reported | 0
Evaluable Treatment Day Baseline Count [Count of Participants; unit: Participants] — indicator for subjects with average treatment day baseline counts greater than or equal to 3.0 log10 colony forming units (CFU)/cm^2 on the 3 test sites (center, mid-peripheral and peripheral) in the treatment area.
  Participants
    Evaluable Subjects | 20
    Non-evaluable Subjects | 8

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Log Change of Skin Flora Relative to Pre-treatment (Baseline) in Each of 3 Sampling Sites at a Defined Post-treatment Sampling Time.
Description: The primary measure of efficacy is change in skin flora log10 CFU/cm^2 in each of the skin sampling sites relative to baseline skin flora log10 CFU/cm^2. Baseline samples must satisfy the greater than or equal to 3.0 in each of the sampling sites, to be used for data analysis.
Time Frame: Post-treatment sampling randomized as 10-minute or 13-minute post-product application
Population: The primary analysis data set used a Modified Intent to Treat population: Subjects were excluded who did not meet the baseline requirement of greater than or equal to 3.0 log10 CFU/cm2 in all three sampling sites on the treatment site. The sampling time for efficacy evaluation was 10 minutes or 13 minutes post-product application as per the randomization schedule.
Measure: Mean (Standard Deviation); unit: log10 CFU/cm^2
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG /IPA Prep - Mid-peripheral: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; sample collected from mid-peripheral test site on skin in application area.
- 3M CHG/IPA Prep - Peripheral: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; sample collected from peripheral test site on skin in application area.
Arm/Group | 3M CHG/IPA Prep / Center | 3M CHG /IPA Prep - Mid-peripheral | 3M CHG/IPA Prep - Peripheral
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (test sites on skin) | 20 | 20 | 20
log10 CFU/cm^2 | -2.19 (1.31) | -1.85 (1.57) | -2.42 (1.20)
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep / Center; Test type: Other — Mixed Model ANOVA with subject as a random effect; p = 0.34, ANOVA — F test

2. Other Pre Specified Outcome: Safety Outcome Evaluated by Skin Irritation Assessment
Description: Skin irritation (dryness, edema, erythema, rash) assessed on the test sites using a 0-3 rating scale: 0 = no reaction, 1 = mild reaction, 2 = moderate reaction, 3 = severe reaction.
Time Frame: Assessed pre-treatment (baseline) and post-treatment (10 or 13 minutes)
Population: All treated subjects were considered evaluable for safety. Safety assessments were based on evaluations for skin reactions at the test sites.
Measure: Number; unit: participants
Arm/Group | 3M CHG/IPA Prep / Center | 3M CHG/IPA Prep / Mid-peripheral | 3M CHG/IPA Prep - Peripheral
Number analyzed (Participants) | 28 | 28 | 28
participants
  Dryness - pre-treatment rating = 0 | 28 | 28 | 28
  Dryness - post-treatment rating = 0 | 28 | 28 | 28
  Edema - pre-treatment rating = 0 | 28 | 28 | 28
  Edema - post-treatment rating = 0 | 28 | 28 | 28
  Erythema - pre-treatment rating = 0 | 28 | 28 | 28
  Erythema - post-treatment rating = 0 | 28 | 28 | 28
  Rash - pre-treatment rating = 0 | 28 | 28 | 28
  Rash - post-treatment rating = 0 | 28 | 28 | 28

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the treatment phase of the study. Treatment procedures required approximately 1 hour for each subject on the test day, and product remained on each subject's skin for approximately 13 to 16 minutes.
Groups:
- 3M CHG/IPA Mid-peripheral: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; sample collected from mid-peripheral test site on skin in application area.
- 3M CHG/IPA Peripheral: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% solution applied topically to intact skin; sample collected from peripheral test site on skin in application area.
Arm/Group | 3M CHG/IPA Prep / Center | 3M CHG/IPA Mid-peripheral | 3M CHG/IPA Peripheral
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03681990/Prot_SAP_000.pdf